CLINICAL TRIAL: NCT00366145
Title: A Phase III, Randomized, Double Blind, Placebo-Controlled Study to Evaluate the Efficacy and Safety of Prochymal® (Ex-vivo Cultured Adult Human Mesenchymal Stem Cells) Infusion for the Treatment of Patients Who Have Failed to Respond to Steroid Treatment for Acute GVHD
Brief Title: Efficacy and Safety of Adult Human Mesenchymal Stem Cells to Treat Steroid Refractory Acute Graft Versus Host Disease (GVHD)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Mesoblast, Inc. (Industry)
Responsible Party: Sponsor
Organization: Mesoblast, Ltd. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 280; NCT00476840 (obsolete NCT alias)
Record Dates: First submitted 2006-08-17; First posted 2006-08-21 (Estimated); Last update posted 2022-02-10 (Actual); Status verified 2022-02

CONDITIONS: Graft Versus Host Disease
Keywords: Acute GVHD; Steroid refractory GVHD; Severe steroid refractory acute GVHD; Steroid refractory; Steroid Refractory Acute Graft Versus Host Disease
MeSH Terms: conditions — Graft vs Host Disease | interventions — remestemcel-l; Excipients; Standard of Care

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Prochymal® (Active Comparator): Participants who receive standard of care plus treatment with ex vivo cultured adult human mesenchymal stem cells.
  Interventions: Biological: Prochymal®; Drug: Standard of Care for GVHD
- Placebo (Placebo Comparator): Participants who receive standard of care and do not receive treatment with ex vivo cultured adult human mesenchymal stem cells.
  Interventions: Drug: Placebo; Drug: Standard of Care for GVHD

INTERVENTIONS:
Biological: Prochymal® — 2 infusions of 2 million cells/kg per week for 4 weeks
  Other Names: Mesenchymal Stem Cells
  Arms: Prochymal®
Drug: Placebo — 2 infusions per week for 4 weeks
  Other Names: excipients without adult human mesenchymal stem cells
  Arms: Placebo
Drug: Standard of Care for GVHD — Institutionally defined standard of care (e.g., maintenance of steroid treatment and the addition of a second-line therapy)

SUMMARY:
The purpose of this study is to evaluate the efficacy and gather additional safety information for Prochymal® in participants who have failed to respond to steroid treatment of Grades B-D acute GVHD.

DETAILED DESCRIPTION:
Approximately 6300 patients receive allogeneic hematopoietic stem cell transplants in the United States each year (International Bone Marrow Transplant Registry [IBMTR], 2003). Nearly 50% (approximately 3,150) of these patients develop acute GVHD (Goker et al). A fraction of these patients (approximately 870) will progress to the severe stages of the disease, Grades III-IV. It is estimated that nearly 82% of those patients with severe acute GVHD will be steroid refractory (Przepiorka et al., 1995) and of these, only 50% of steroid-refractory patients will respond to secondary and tertiary treatments (Greinix et al., 2000). Thus, roughly 350 patients each year face tremendous odds against survival. In addition, most patients who initially responded to secondary and tertiary treatments have a high risk of dying within the first year (Remberger et al., 2001; Anasetti et al., 1994). Development of new therapeutic agents and strategies to rescue patients with steroid refractory, acute GVHD would provide a significant benefit in an area of unmet medical need. Participants will receive standard of care in addition to adult mesenchymal stem cells or placebo.

ELIGIBILITY:
Inclusion Criteria:

* Participant must be 6 months to 70 years of age, inclusive.
* Participants who have failed to respond to steroid treatment.

Failure to respond to steroid treatment is defined as any grade B-D (IBMTR) grading of acute GVHD that shows:

* No improvement after 3 days and a duration of no greater than 2 weeks while receiving treatment with methylprednisolone (greater than or equal to 1 mg/kg/day) or equivalent.
* Participant must be treated within 4 days of randomization. In urgent situations 2nd line therapy may be started 24 hours prior to randomization, and Prochymal® must be initiated within the following 3 days.
* Participants who have received an increase in their steroid dose treatment prior to randomization will be eligible for enrollment. An increase in steroid dose will not be considered as second line therapy.
* Participant must have adequate renal function as defined by: Calculated Creatinine Clearance of >30 milliliters per minute (mL/min) using the Cockcroft-Gault equation.
* For pediatric participants: Schwartz equation: (Participant population: infants over 1 week old through adolescence (<18 years old).
* Participants who are women of childbearing potential must be non-pregnant, not breast-feeding, and use adequate contraception. Male participants must use adequate contraception.
* Participant must have a minimum Karnofsky Performance Level of at least 30 at the time of study entry.
* Participant (or legal representative where appropriate) must be capable of providing written informed consent.

Exclusion Criteria:

* Participant has started treatment with second line therapy >24 hours prior to randomization.
* Participant has received agents other than steroids for primary treatment of acute GVHD.
* Participant is participating in the CTN Protocol 0302.
* Participant has any underlying or current medical or psychiatric condition that, in the opinion of the Investigator, would interfere with the evaluation of the participant including uncontrolled infection, heart failure, pulmonary hypertension, etc.
* Participant may not receive any other investigational agents (not approved by the FDA) concurrently during study participation or within 30 days of randomization.
* Participant has a known allergy to bovine or porcine products.
* Participant has received a transplant for a solid tumor disease.

Ages: 6 Months to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 260 (Actual)
Dates: Start 2006-08-17 (Actual); Primary Completion 2008-12-26 (Actual); Study Completion 2009-05-28 (Actual)

PRIMARY OUTCOMES:
Percentage of Participants achieving Complete Response of Greater Than or Equal to 28 Days Duration | up to 100 Days post first infusion
  A complete response was defined as complete resolution of all clinical signs of Graft versus host disease (GVHD)- that had to be maintained for at least 28 consecutive days (durable complete response [DCR]) within 100 days post first infusion.

SECONDARY OUTCOMES:
Overall Survival at 180 days Post First Infusion | Day 180
  Percentage of participants who survived at 180 days post first infusion.

CONTACTS AND LOCATIONS:
Overall Officials: Christopher James, PA, Study Director — Mesoblast, Inc.
Locations (70):
- United States (47):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Arizona Cancer Center, Tucson, Arizona
  - City of Hope, Duarte, California
  - Univeristy of California San Francisco, San Francisco, California
  - Yale New Haven Hospital, New Haven, Connecticut
  - University of Miami, Miami, Florida
  - All Children's Hospital, St. Petersburg, Florida
  - Emory University, Atlanta, Georgia
  - Northside Hospital, Atlanta, Georgia
  - Northwestern Center for Clinical Research, Chicago, Illinois
  - Rush University Medical Center, Chicago, Illinois
  - University of Illinois - Chicago, Chicago, Illinois
  - Indiana Blood and Bone Marrow Transplant Center, Beech Grove, Indiana
  - Univeristy of Iowa Hospitals and Clinics, Iowa City, Iowa
  - University of Kansas Medical Center, Kansas City, Kansas
  - University of Louisville, Louisville, Kentucky
  - Louisiana State University, Shreveport, Louisiana
  - University of Maryland/Greenbaum, Baltimore, Maryland
  - Tufts-New England Medical Center, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Karmanos/Wayne State University, Detroit, Michigan
  - Mayo Clinic Rochester, Rochester, Minnesota
  - Univeristy of Mississippi Medical Center, Jackson, Mississippi
  - University of Nebraska, Omaha, Nebraska
  - Hackensack University Medical Center, Hackensack, New Jersey
  - Roswell Park, Buffalo, New York
  - New York Presbyterian Hospital, New York, New York
  - Mount Sinai Medical Center, New York, New York
  - Columbia University/New York Presbyterian Hospital, New York, New York
  - University of Rochester, Rochester, New York
  - New York Medical College, Valhalla, New York
  - Duke University, Durham, North Carolina
  - Wake Forest Univeristy School of Medicine, Winston-Salem, North Carolina
  - Oregon Health and Science University, Portland, Oregon
  - Penn State Hershey Medical Center, Hershey, Pennsylvania
  - Western Pennsylvania Cancer Institute, Pittsburgh, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
  - Texas Cancer Center at Medical City, Dallas, Texas
  - Baylor University, Dallas, Texas
  - Univeristy of Texas Southwestern Medical Center, Dallas, Texas
  - MD Anderson Cancer Center, Houston, Texas
  - Texas Research Center, San Antonio, Texas
  - Virginia Commonwealth/Massey Cancer Center, Richmond, Virginia
  - Fred Hutchinson Cancer Research Center, Seattle, Washington
  - University of Wisconsin Madison, Madison, Wisconsin
  - Medical College of Wisconsin, Milwaukee, Wisconsin
- Australia (3):
  - Royal Brisbane Hospital, Herston, Queensland
  - Royal Melbourne Hospital, Parkville, Victoria
  - Royal Perth Hospital, Perth, Western Australia
- Canada (12):
  - Co-Medica Research Network, Calgary, Alberta
  - British Columbia's Children's Hospital, Vancouver, British Columbia
  - Cancer Care Manitoba, Winnipeg, Manitoba
  - Queen Elizabeth II Health Sciences Centre, Halifax, Nova Scotia
  - Hamilton Health Sciences Centre, Hamilton, Ontario
  - London Health Sciences Centre- Westminster Campus, London, Ontario
  - Ottawa Hospital, Ottawa, Ontario
  - Toronto General Hospital, Toronto, Ontario
  - Princess Margaret Hospital, Toronto, Ontario
  - Maisonneuve-Rosemont Hospital, Montreal, Quebec
  - Hopital Enfant-Jesus, Québec
  - Hopital du Saint-Sacrement, Québec
- Italy (2):
  - Universia degli Studi di Pesaro, Pesaro, PU
  - IRCCS Policlinico San Matteo, Pavia
- Kantonsspital Basel, Basel, Switzerland
- United Kingdom (5):
  - Barts & London School of Medicine, London, England
  - John Radcliffe Hospital, Headington, Oxford
  - Bristol Royal Hospital for Children, Bristol, UK
  - Glasgow Royal Infirmary, Glasgow, UK
  - Leeds General Infirmary, Leeds, UK

REFERENCES:
- [Background] Bartholomew A, Sturgeon C, Siatskas M, Ferrer K, McIntosh K, Patil S, Hardy W, Devine S, Ucker D, Deans R, Moseley A, Hoffman R. Mesenchymal stem cells suppress lymphocyte proliferation in vitro and prolong skin graft survival in vivo. Exp Hematol. 2002 Jan;30(1):42-8. doi: 10.1016/s0301-472x(01)00769-x. PMID 11823036
- [Background] Deans RJ, Moseley AB. Mesenchymal stem cells: biology and potential clinical uses. Exp Hematol. 2000 Aug;28(8):875-84. doi: 10.1016/s0301-472x(00)00482-3. PMID 10989188
- [Background] Lazarus HM, Koc ON, Devine SM, Curtin P, Maziarz RT, Holland HK, Shpall EJ, McCarthy P, Atkinson K, Cooper BW, Gerson SL, Laughlin MJ, Loberiza FR Jr, Moseley AB, Bacigalupo A. Cotransplantation of HLA-identical sibling culture-expanded mesenchymal stem cells and hematopoietic stem cells in hematologic malignancy patients. Biol Blood Marrow Transplant. 2005 May;11(5):389-98. doi: 10.1016/j.bbmt.2005.02.001. PMID 15846293
- [Background] Le Blanc K, Rasmusson I, Sundberg B, Gotherstrom C, Hassan M, Uzunel M, Ringden O. Treatment of severe acute graft-versus-host disease with third party haploidentical mesenchymal stem cells. Lancet. 2004 May 1;363(9419):1439-41. doi: 10.1016/S0140-6736(04)16104-7. PMID 15121408
- [Background] Le Blanc K, Pittenger M. Mesenchymal stem cells: progress toward promise. Cytotherapy. 2005;7(1):36-45. doi: 10.1080/14653240510018118. PMID 16040382
- [Derived] Camilleri ET, Gustafson MP, Dudakovic A, Riester SM, Garces CG, Paradise CR, Takai H, Karperien M, Cool S, Sampen HJ, Larson AN, Qu W, Smith J, Dietz AB, van Wijnen AJ. Identification and validation of multiple cell surface markers of clinical-grade adipose-derived mesenchymal stromal cells as novel release criteria for good manufacturing practice-compliant production. Stem Cell Res Ther. 2016 Aug 11;7(1):107. doi: 10.1186/s13287-016-0370-8. PMID 27515308
- See also: Description Click here for more information about this study: A Phase III Study to Evaluate the Efficacy and Safety of Prochymal® (Ex vivo Cultured Adult Human Mesenchymal Stem Cells) Infusion for the Treatment of Steroid-Refractory Acute GVHD — http://www.osiris.com